CLINICAL TRIAL: NCT05458700
Title: POS-cUTI:Perpetual Observational Study on Complicated Urinary Tract Infections
Brief Title: POS-cUTI: Study on Complicated Urinary Tract Infections
Status: Recruiting | Type: Observational
Sponsor: European Clinical Research Alliance for Infectious Diseases (ECRAID) (Other)
Collaborators: UMC Utrecht (Other); Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: ECRAID-Base POS-cUTI
Record Dates: First submitted 2022-05-20; First posted 2022-07-14 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Urinary Tract Infections
Keywords: UTI; European clinical research network; Randomized ITUs research activities
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: None Retained — Urine culture, blood culture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collect information — Collect information from the patients to support the design of innovate clinical trials

SUMMARY:
Urinary tract infections (UTI) are among the most common infectious diseases and the most frequent source of community, healthcare-associated and nosocomial bacteraemia. They are associated with significant morbidity and mortality. Due to the high frequency of UTI, they have a major impact on antibiotic use and the antimicrobial resistance of prominent UTI pathogens is of recognised importance. Therefore, UTIs, and particularly complicated urinary tract infections cUTIs, are a target for repurposing of old and neglected drugs, new drug development and non-antibiotic therapeutic and preventive approaches.

ELIGIBILITY:
Inclusion Criteria:

* A documented microbial pathogen on culture of blood OR urine according to standards of interpretation regarding to the type of infection, pathogen, quantitative culture results and sample. Guide for adequate interpretation is detailed in Lab Manual. However, if the local laboratory uses diferent microbiological criteria, patients will be elegible and the criteria used will be collected AND
* Local and systemic signs and symptoms of UTI including at least one of these two: (a) fever (i.e.,temperature greater than 38ºC), chills or malaise; and (b) flank pain, back pain, costo-vertebral angle pain or tenderness, dysuria or urinary urgency, AND
* It occurs in the presence of a functional or anatomical abnormality of the urinary tract or in the presence of catheterization, including (but not limited to) presence of a urinary catheter; 100 mL or more of residual urine after voiding (neurogenic bladder); obstructive uropathy (nephrolithiasis, fibrosis); azotemia caused by intrinsic renal disease; urinary retention, including retention caused by benign prostatic hypertrophy.
* Patients with pyelonephritis or bacteremia with a urinary tract source, regardless of underlying abnormalities of the urinary tract, are also to be included.
* Patients with urinary catheter presenting with fever, bacteriuria and bacteraemia caused by the same urinary pathogen can be included if other sources of bacteraemia are reasonably discarded.
* Depending on the country regulation: The patient, family or legally authorised representative signed the informed consent to participate or; notification of non-objection to the use of pseudo-anonymized personal and medical data.

Exclusion Criteria:

* Patients with a life expectancy previous to development of cUTI <30 days and those exclusively under palliative care in whom any eventually needed invasive procedure would not be performed.
* Patients who died in <48 hours since the presentation with cUTI
* Patients participating in RCT for treatment of cUTI
* >96 hours since from the clinical diagnosis of cUTI. I.e. >96 hours from positive urine/blood culture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) patients admitted to an acute care hospital with cUTI, or developing cUTI during hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To delineate the outcomes of patients with cUTI, and the impact of managemnt-related variables; specifically the incidence of treatment failure in patients with cUTI and modifiable and non-modifiable risk factors for treatment failure | 4 years
  Clinical and microbiological cure at test of cure (TOC; 14-21 days ±3 days after the diagnosis of cUTI).
  Clinical cure is defined as the resolution of all new signs and symptoms related to cUTI and no need to continue with antibiotics; microbiological cure requires urine culture with <103 CFU/mL of the initial pathogen. Whenever clinical and microbiological cure at TOC is not reached, it will be considered as failure.

SECONDARY OUTCOMES:
To describe the patient population with cUTI and the microbiological aetiology of cUTI in the study sites. | 4 years
  Urine culture indicative of cUTI: performed/not, date, positive/negative, if positive: micoorganism, susceptibility. Date of susceptibility report
To determine the rate of recurrences and superinfections, and those caused by multidrugresistant organisms | 4 years
  Recurrence of UTI (relapses and reinfections) in the first 30 days follow-up. Recurrence is defined as the reappearance of symptoms of urinary tract infection together with a positive blood culture or urine culture for the same microorganism isolated in the initial blood culture after having reached clinical and microbiological cure. Reinfection is defined in a similar way. Superinfections are other infections different from UTI.
  but with isolation of a bacteria or strain different from the initial one. Superinfections other infections different from UTI)
To determine the mortality and its predictors in patients with cUTI. | 4 years
  All-cause 30-day mortality
To determine the length of hospital stay after cUTI | 4 years
  Hospital stay after index cUTI episode in days.
To describe variations in current practices in treating cUTI in the study sites. | 4 years
  Type of acquisition, urine culture indicative of cUTI, blood culture at days 0 and , location of cUTI, purulent complications, radiological and blood and urine test data, Pitt and SOFA scores, severity of systemic response, treatment of infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: No